CLINICAL TRIAL: NCT03062189
Title: Binge Drinking Among Young Students is a Risk Factor for the Development of Alcohol Use Disorders: Results From an Epidemiologic-observational Study
Brief Title: Binge Drinking Among Youngs is a Risk Factor for Alcohol Use Disorders
Status: Completed | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Giovanni Addolorato, Principal Investigator, Catholic University of the Sacred Heart
Other Study IDs: BingeDrinkingamongYoungStudy
Record Dates: First submitted 2016-12-14; First posted 2017-02-23 (Actual); Last update posted 2017-02-27 (Actual); Status verified 2017-01

CONDITIONS: Binge Drinking
MeSH Terms: conditions — Binge Drinking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study was to assess drinking habits and patterns of alcohol consumption, smoking habits, use of illicit drugs and the prevalence of binge drinking and alcohol use disorders among Italian young students. Furthermore to investigate the correlation between binge drinking and alcohol use disorders.

DETAILED DESCRIPTION:
This study was performed on 2,704 subjects attending high school, through the administration of questionnaires regarding socio-demographic data, anthropometric characteristics, pattern and amount of alcohol intake, smoking habits, use of illicit drugs and physical activity were administered to students. Moreover mood and anxiety were evaluated through AUDIT, STAI-Y1, STAY-Y2 and ZUNG. The aim of the study was to assess drinking habits and patterns of alcohol consumption, smoking habits, use of illicit drugs and the prevalence of binge drinking and alcohol use disorders among Italian young students. Furthermore to investigate the correlation between binge drinking and alcohol use disorders.

ELIGIBILITY:
Inclusion Criteria:

* Subjects attending high school of three italian cities (Rome, Latina, Frosinone)
* Subjects aged between 13 and 19 years
* Subjects that accept the interview

Exclusion Criteria:

* Subjects that don't accept the interview

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 2,704 subjects attending high school in three italian cities
Sampling Method: Probability Sample
Enrollment: 2704 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Binge drinking behavior | 1 year
  Binge drinking behavior was defined as an alcohol consumption of more than 5 drinks within about two hour period

SECONDARY OUTCOMES:
Amount of alcoholic beverage consumed | 1 year
  One drink is defined as an amount of alcoholic beverages containing 12 g of absolute alcoho
Type of alcoholic beverage consumed | 1 year
Frequency of alcohol consumption | 1 year
Alcohol consumption outside meals | 1 year
  One drink is defined as an amount of alcoholic beverages containing 12 g of absolute alcoho
Frequency of alcohol drinking outside meals | 1 year
  One drink is defined as an amount of alcoholic beverages containing 12 g of absolute alcoho
Amount of cigarettes smoked | 1 year
Frequency of cigarettes smoked | 1 year
Type of illicit drugs used | 1 year
Frequency of illicit drugs used | 1 year
Diagnosis of Alcohol Use Disorder | 1 year
  According AUDIT score
STAI score | 1 year
  STAI assess existing anxiety a predisposition to anxious reaction as a personality characteristic. Itis structuredby two axes (y1 for state anxiety and y2 for trait anxiety), both consisting of 20 multiple-choice items; each item has a score from 1 to 4; the total score of y1 and y 2 axes can range from 20 to 80. This test was selected for simplicity, validity and reliability. The subjects evaluated were divided as high and low anxious and a value of 40 was used to distinguish the two groups
Zung-SDS | 1 year
  Zung-SDS constitutes an effective instrument in screening for depression and its positive predictive value of a diagnosis of depression is between 88.7% and 92.3%. The Zung-SDS contains 20 multiple items with a score from 1 to 4 each; total score above 50 indicates a condition of depression

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Addolorato, MD, Principal Investigator — Catholic University of Sacred Heart, Rome

IPD SHARING:
Plan to Share IPD: No